CLINICAL TRIAL: NCT02586012
Title: Weight-based Dosing in Hemophilia A: A Randomized, Controlled, Open-label, Crossover Trial to Measure Factor VIII Recovery Following Factor VIII Concentrate Dosing Based on Total Body Weight, Ideal Body Weight, and Lean Body Mass
Brief Title: Weight-based Dosing in Hemophilia A
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Craig Seaman (Other)
Responsible Party: Sponsor-Investigator, Craig Seaman, Assistant Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PRO15010061
Record Dates: First submitted 2015-10-22; First posted 2015-10-26 (Estimated); Results first posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; factor VIII-Fc fusion protein; F8 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- TBW, LBM, IBW (Experimental): Subjects will be randomized to receive rFVIII doses calculated by 3 separate methods over a 3 week period. Week 1, the dose will be based on TBW (Total Body Weight); Week 2, the dose will be based on LBM (Lean Body Mass); and Week 3, the dose will be based on IBW (Ideal Body Weight).
  Interventions: Drug: rFVIII
- LBM, IBW, TBW (Experimental): Subjects will be randomized to receive rFVIII doses calculated by 3 separate methods over a 3 week period. Week 1, the dose will be based on LBM (Lean Body Mass); Week 2, the dose will be based on IBW (Ideal Body Weight); and Week 3, the dose will be based on TBW (Total Body Weight).
  Interventions: Drug: rFVIII
- IBW, TBW, LBM (Experimental): Subjects will be randomized to receive rFVIII doses calculated by 3 separate methods over a 3 week period. Week 1, the dose will be based on IBW (Ideal Body Weight); Week 2, the dose will be based on TBW (Total Body Weight); and Week 3, the dose will be based on LBM (Lean Body Mass).
  Interventions: Drug: rFVIII
- TBW, IBW, LBM (Experimental): Subjects will be randomized to receive rFVIII doses calculated by 3 separate methods over a 3 week period. Week 1, the dose will be based on TBW (Total Body Weight); Week 2, the dose will be based on IBW (Ideal Body Weight); and Week 3, the dose will be based on LBM (Lean Body Mass).
  Interventions: Drug: rFVIII
- LBM, TBW, IBW (Experimental): Subjects will be randomized to receive rFVIII doses calculated by 3 separate methods over a 3 week period. Week 1, the dose will be based on LBM (Lean Body Mass); Week 2, the dose will be based on TBW (Total Body Weight); and Week 3, the dose will be based on IBW (Ideal Body Weight).
  Interventions: Drug: rFVIII
- IBW, LBM, TBW (Experimental): Subjects will be randomized to receive rFVIII doses calculated by 3 separate methods over a 3 week period. Week 1, the dose will be based on, IBW (Ideal Body Weight); Week 2, the dose will be based on LBM (Lean Body Mass); and Week 3, the dose will be based on TBW (Total Body Weight).
  Interventions: Drug: rFVIII

INTERVENTIONS:
Drug: rFVIII — Recombinant FVIII concentrate is an FDA approved, and both efficacious and safe, therapy for the treatment and prevention of bleeding in hemophilia A. The rFVIII infusion dose will be calculated as follows: [(weight in kg x desired FVIII increase of 100 IU/dL)/(2)].
  Other Names: eloctate, advate, helixate, kogenate, recombinant

SUMMARY:
Hemophilia A is an inherited (genetic) disease where a protein, factor VIII (FVIII), which promotes blood clotting is missing or does not work properly. Individuals with hemophilia A are at risk for bleeding. Bleeding is prevented and/or treated with recombinant factor VIII (rFVIII), which is an FDA-approved treatment for Hemophilia A. Obesity is common among patients with hemophilia. Some studies have shown that obese hemophilia patients may be able to prevent bleeding with a lower dose of clotting factor than the dose they are currently receiving. The lower dose is calculated based on what a patient should weigh rather than what he does weigh. This is a clinical research study to test whether calculating rFVIII dosing based on lean body mass and ideal body weight (what a person should weigh based on his height) in overweight and obese patients with hemophilia is more accurate than calculating rFVIII dosing based on what a person actually weighs.

DETAILED DESCRIPTION:
The investigators propose a single center, randomized, controlled, open-label, crossover trial to determine if recombinant factor VIII (rFVIII) dosed according to lean body mass (LBM) and ideal body weight (IBW) achieves a targeted FVIII recovery with better precision than based on total body weight (TBW). The investigators hypothesize the use of LBM and IBW to determine the dose of rFVIII necessary to attain a desired FVIII recovery of 2 +/- 0.2 IU/dl per IU/kg (100 +/- 10%) in overweight and obese (body mass index greater than or equal to 25 mg/m2), adult males (age 18 or older) with hemophilia A (FVIII activity 40% or less) will result in a 50% greater proportion of subjects within this range when compared to TBW. Eligible patients receiving care at the Hemophilia Center of Western Pennsylvania (HCWP) will be enrolled during clinic visits. Following enrollment and completion of screening assessment, subjects will present to HCWP for three study visits with each study visit occurring on successive weeks. Subjects will not have received any rFVIII for a period of at least 72 hours prior to each study visit. Recombinant FVIII infusion based on TBW, LBM, or IBW will take place during each study visit, and the order will be determined by randomization. During each study visit, FVIII levels will be assessed by obtaining blood samples before and at 10 and 30 minutes and 1 hour after infusion. Outcomes include the proportion of subjects achieving a desired peak FVIII recovery value of 2 +/- 0.2 IU/dl per IU/kg (100 +/- 10%) at 10 minutes following infusion of rFVIII dosed according to LBM and TBW, IBW and TBW, and LBM and IBW. The investigators will use mixed effects logistic regression to investigate the effect of using different weight-based dosing methods on attaining target FVIII levels. We aim to have 24 subjects successfully complete the study.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males age 18 or older.
2. Hemophilia A (FVIII activity 40% or less).
3. Overweight or obesity defined as a BMI of 25.0-29.9 and ≥ 30 mg/m2, respectively.

Exclusion Criteria:

1. Prior history of, or currently detectable, FVIII inhibitor defined as greater than or equal to 0.6 Bethesda Units (BU); however, a subject with a past low-level non-responding inhibitor defined as less than 5 BU, with no increase in titer following FVIII exposure, and not detectable within 12 months of the study, despite FVIII exposure during that period, will be allowed to enroll on study.
2. Allergy to FVIII products.
3. Current rFVIII requirements do not include at least a 72-hour period without rFVIII administration.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Seaman, MD, MS, Principal Investigator — University of Pittsburgh
Locations (1):
- Hemophilia Center of Western Pennsylvania, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TBW, LBM, IBW | LBM, IBW, TBW | IBW, TBW, LBM | TBW, IBW, LBM | LBM, TBW, IBW | IBW, LBM, TBW
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 4 | 2 | 4 | 3 | 4 | 2
Not Completed | 1 | 3 | 1 | 2 | 1 | 3
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 1 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1
Not completed — study terminated | 0 | 2 | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Subjects: All subjects randomized to 1 of 6 possible dosing sequence scenarios based on 3 different weight-based dosing regimens (TBW, LBM, and IBW).
Arm/Group | Subjects
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.6 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: cm] | 178.5 (6.9)
Weight [Mean (Standard Deviation); unit: kg] | 93.0 (13.6)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.2 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Dosed Based on LBM (Lean Body Mass) and TBW (Total Body Weight) Achieving Desired Peak FVIII Recovery.
Description: Desired peak FVIII recovery value of 2 +/- 0.2 IU/dl per IU/kg (100 +/- 10%) at 10 minutes following infusion based on LBM and TBW. FVIII recovery values will be calculated as follows: [(weight in kg x observed FVIII recovery in IU/dL)/(dose in IU)] and expressed as IU/dL per IU/kg.
Time Frame: 3 weeks
Population: Subjects receiving rFVIII based on LBM and TBW.
Measure: Count of Participants; unit: Participants
Groups:
- Lean Body Mass: Subjects receiving rFVIII based on LBM.
- Total Body Weight: Subjects receiving rFVIII based on TBW.
Arm/Group | Lean Body Mass | Total Body Weight
Number analyzed (Participants) | 20 | 20
Participants | 9 | 6
Statistical Analysis 1: Comparison: Lean Body Mass vs Total Body Weight; Test type: Superiority; p < 0.05, Mixed Models Analysis

2. Secondary Outcome: Proportion of Subjects Dosed Based on IBW (Ideal Body Weight) and TBW (Total Body Weight) Achieving Desired Peak FVIII Recovery.
Description: Desired peak FVIII recovery value of 2 +/- 0.2 IU/dl per IU/kg (100 +/- 10%) at 10 minutes following infusion based on IBW and TBW. FVIII recovery values will be calculated as follows: [(weight in kg x observed FVIII recovery in IU/dL)/(dose in IU)] and expressed as IU/dL per IU/kg.
Time Frame: 3 weeks
Population: Subjects receiving rFVIII based on IBW and TBW.
Measure: Count of Participants; unit: Participants
Groups:
- Ideal Body Weight: Subjects receiving rFVIII based on IBW.
Arm/Group | Ideal Body Weight | Total Body Weight
Number analyzed (Participants) | 20 | 20
Participants | 10 | 6
Statistical Analysis 1: Comparison: Ideal Body Weight vs Total Body Weight; Test type: Superiority; p < 0.05, Mixed Models Analysis

3. Secondary Outcome: Proportion of Subjects Dosed Based on LBM (Lean Body Mass) and IBW (Ideal Body Weight) Achieving Desired Peak FVIII Recovery.
Description: Desired peak FVIII recovery value of 2 +/- 0.2 IU/dl per IU/kg (100 +/- 10%) at 10 minutes following infusion based on LBM and IBW. FVIII recovery values will be calculated as follows: [(weight in kg x observed FVIII recovery in IU/dL)/(dose in IU)] and expressed as IU/dL per IU/kg.
Time Frame: 3 weeks
Population: Subjects receiving rFVIII based on LBM and IBW.
Measure: Count of Participants; unit: Participants
Arm/Group | Lean Body Mass | Ideal Body Weight
Number analyzed (Participants) | 20 | 20
Participants | 9 | 10
Statistical Analysis 1: Comparison: Lean Body Mass vs Ideal Body Weight; Test type: Superiority; p < 0.05, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 3 weeks
Groups:
- Total Body Weight: Subjects who received rFVIII based on TBW.
- Ideal Body Weight: Subjects who received rFVIII based on IBW.
- Lean Body Mass: Subjects who received rFVIII based on LBM.
Arm/Group | Total Body Weight | Ideal Body Weight | Lean Body Mass
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
Early termination due to poor enrollment prior to 24 subjects successfully completing the study.

The rFVIII dose was erroneously calculated in 7 subjects resulting in the administration of a smaller than intended amount.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/12/NCT02586012/Prot_SAP_000.pdf